CLINICAL TRIAL: NCT02741427
Title: Safety, Acceptability and Efficacy of a Silica Dentifrice Containing Blue Pigment on Tooth Whitening: a Randomized Clinical Trial
Brief Title: Efficacy of a Whitening Dentifrice on Tooth Discoloration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Principal Investigator, Jossaria Pereira de Sousa, Master degree in Dentistry, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUofParabia
Record Dates: First submitted 2016-04-11; First posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Tooth Discoloration
Keywords: Tooth discoloration; Toothpaste; Tooth bleaching; Clinical trial
MeSH Terms: conditions — Tooth Discoloration | interventions — hydrated silica gel-based toothpaste; Carbamide Peroxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- G1 (group 1) - Conventional toothpaste (Placebo Comparator): G1 used a conventional toothpaste in daily oral regimen
  Interventions: Other: Conventional toothpaste
- G2 (group 2) - Whitening toothpaste (Experimental): G2 used a whitening toothpaste containing blue pigment in daily oral regimen
  Interventions: Other: Whitening toothpaste
- G3 (group 3) - 10 % Carbamide peroxide (Active Comparator): G3 made an at-home tooth bleaching with 10 % Carbamide peroxide
  Interventions: Other: 10% carbamide peroxide

INTERVENTIONS:
Other: Conventional toothpaste — The participants should brush their teeth with conventional toothpaste for 90 seconds, twice per day, during two weeks.They should place a pea-size amount of toothpaste on their toothbrushes, use dental floss, but not mouth rinse.
  Other Names: Colgate Máxima Proteção Anticáries
  Arms: G1 (group 1) - Conventional toothpaste
Other: Whitening toothpaste — The subjects should brush teeth with whitening toothpaste containing blue pigment for 90 seconds, twice per day, during two weeks.They should place a pea-size amount of toothpaste on toothbrushes, use dental floss, but not mouth rinse.
  Other Names: Close up White Now
  Arms: G2 (group 2) - Whitening toothpaste
Other: 10% carbamide peroxide — The subjects should dispense the bleaching gel at night into the trays (maxillary and mandibular) and to insert them to cover at least the anterior teeth for a period of 4 h per day, over a 2-week period. Both arches should be bleached at the same time. During the period of bleaching, volunteers should receive the same toothpaste used by G1, in other words, without "whitening agents", to standardize their oral hygiene regimen
  Other Names: Whiteness perfect 10%
  Arms: G3 (group 3) - 10 % Carbamide peroxide

SUMMARY:
The purpose of this study was to compare the whitening effect of a toothpaste containing blue pigment with a conventional toothpaste and with at-home tooth bleaching; evaluate the subject's perception about tooth color improvement and; and evaluate the safety and acceptability of these products.

DETAILED DESCRIPTION:
The study was approved by local Ethical Committee under protocol number CAAE: 035541412.7.0000.5188, and each volunteer signed an informed consent form prior to enrollment in the study.

The sample size calculation was carried out based on a previous study. To detect the bleaching effect with a power of 80% and a one-tailed alpha error of 5%, a sample size of 20 subjects in each treatment group was necessary to detect a 20% difference between groups in shade change. A 20% addiction in subjects' number, taking into consideration potential loss or refusal, gave a total sample size of 75 subjects (25 in each group). The individuals were invited to participate in this clinical trial through advertisement exposed at the Federal University of Paraíba, Brazil.

Basing on eligibility criteria, 75 volunteers were selected to the trial and randomized to one of the three groups of treatment: G1- brushing teeth with a conventional toothpaste; G2- brushing teeth with a silica whitening dentifrice containing blue pigment; and G3 - at-home tooth bleaching with 10% carbamide peroxide. The treatments will be detailed in another section. It was used a simple randomization to allocate the subjects, and a randomization table was prepared in the Excel Program by a member, not directly involved with the clinical part of the study.

To mask the products used in the treatment groups, each toothpaste type was enveloped with an adhesive tape of a different color and the seal of the bleaching gel syringe was removed. The same examiner responsible for subject allocation did this procedure. Thus, testing with the toothpastes was double-blinded, where both evaluator and subject did not know which toothpaste was being used.

The outcomes evaluated were: tooth shade, subjects' perception about tooth color appearance, and safety and acceptability of products tested, which were measured at baseline, 2-weeks, 3-weeks and 4-weeks of the beginning of treatments.

For statistical analysis, data were checked for normal distribution using the Kolmogorov Smirnov test, and then it was applied the appropriated parametric or non-parametric tests. Differences were considered statistically significant when p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* To have six maxillary anterior teeth with a mean shade of C1 or darker (Vitapan Classical, Vita Zahnfabrik, Bad Sackingen, Germany),

Exclusion Criteria:

* With active caries or periodontal disease,
* Presenting non-vital anterior teeth,
* Previous hypersensitivity,
* Under orthodontic treatment,
* With structural defect in the enamel,
* Who had used tooth whiteners within the previous 3 years,
* Smokers,
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Tooth shade changes from baseline until 4 weeks of the beginning of intervention | Baseline, Immediately after first product application, 2 weeks and 4 weeks of the beginning of interventions
  The tooth shade evaluation was performed at each time frame using the digital spectrophotometer that provided tooth shade via two different methods: using the 16 shade tabs in the Vita shade guide (B1-C4); and the CIEL*a*b* color system. The difference between the color coordinates was calculated as: ∆E*= [(∆L*)2 + (∆a*)2 + (∆b*)2]1/2, where ΔL*, Δa*, and Δb* are the mathematical differences among CIE L*, a*, and b* at the different time frames and baseline measurements.

SECONDARY OUTCOMES:
Subjects' perception about improvement on tooth color | 2 weeks of the beginning of interventions
  After two weeks of treatment, the subjects received a visual analog scale (VAS) ranging from 1 (no improvement in tooth appearance) to 7 (exceptional improvement in tooth appearance), in order to evaluate their satisfaction level with tooth appearance
Tooth sensitivity and gingival irritation evaluation | Daily during three weeks
  Each subject should record tooth sensitivity or gingival irritation on a daily basis for 3 weeks (2 weeks of treatment and 1 week after treatment). They should use a standardized grading scale ranked as follows: 0, no sensitivity; 1, mild sensitivity; 2, moderate sensitivity; 3, considerable sensitivity; and 4, severe sensitivity
Acceptability of interventions | 2 weeks of the beginning of interventions
  The acceptability of the three products was assessed using a questionnaire containing six questions about the opinion of subjects regarding the treatment regimen adopted. The questions were scored from positive to negative answers, as follows: 1, agree; 2, neither agree nor disagree; and 3, disagree. The questions related to sufficient instruction, ease of use, comfort level, perceived taste, and overall satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jossaria P Sousa, Master, Principal Investigator — Federal University of Paraiba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meireles SS, Santos IS, Bona AD, Demarco FF. A double-blind randomized clinical trial of two carbamide peroxide tooth bleaching agents: 2-year follow-up. J Dent. 2010 Dec;38(12):956-63. doi: 10.1016/j.jdent.2010.08.003. Epub 2010 Aug 13. PMID 20709137
- [Background] Walsh TF, Rawlinson A, Wildgoose D, Marlow I, Haywood J, Ward JM. Clinical evaluation of the stain removing ability of a whitening dentifrice and stain controlling system. J Dent. 2005 May;33(5):413-8. doi: 10.1016/j.jdent.2004.10.021. Epub 2004 Dec 20. PMID 15833397